CLINICAL TRIAL: NCT04644237
Title: A Phase 2, Multicenter, Randomized Study of Trastuzumab Deruxtecan in Subjects With HER2-mutated Metastatic Non-small Cell Lung Cancer (NSCLC) (DESTINY-LUNG02)
Brief Title: Trastuzumab Deruxtecan in Participants With HER2-mutated Metastatic Non-small Cell Lung Cancer (NSCLC)
Acronym: DESTINY-LUNG02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS8201-A-U206; 2020-003427-42 (EudraCT Number)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Trastuzumab Deruxtecan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan 6.4 mg/kg (Experimental): Participants will be randomized to receive trastuzumab deruxtecan 6.4 mg/kg administered by intravenous infusion every 3 weeks (Q3W).
  Interventions: Drug: Trastuzumab deruxtecan
- Trastuzumab deruxtecan 5.4 mg/kg (Experimental): Participants will be randomized to receive trastuzumab deruxtecan 5.4 mg/kg administered by intravenous infusion every 3 weeks (Q3W).
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan 100 mg will be provided as a sterile lyophilized powder and reconstituted with 5 mL water for injection (final concentration 20 mg/mL [ie, 100 mg/5 mL]). The study drug will be administered as an intravenous (IV) infusion over 30 to 90 min Q3W ± 2 days. The initial dose of study drug will be infused for 90 ± 10 min.

SUMMARY:
This study was designed to evaluate the safety and efficacy of trastuzumab deruxtecan in HER2-mutated metastatic non-small cell lung cancer (NSCLC) participants who had disease recurrence or progression during/after at least one regimen of prior anticancer therapy (second line or later) that must have contained a platinum-based chemotherapy drug.

DETAILED DESCRIPTION:
This randomized, two-arm, phase 2, multicenter study will evaluate the safety and efficacy of 5.4 mg/kg and 6.4 mg/kg trastuzumab deruxtecan administered every 3 weeks (Q3W) in participants with HER2-mutated metastatic NSCLC. Each participant is expected to receive approximately 14 months of trastuzumab deruxtecan treatment. The primary endpoint of the study will be confirmed objective response rate (blinded independent central review). Secondary endpoints will include, but not limited to, disease control rate, duration of response, progression-free survival, objective response rate (investigator), overall survival, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women ≥18 years, follow local regulatory requirements if the legal age of the consent for study participation is >18 years
* Pathologically documented metastatic NSCLC with a known activating HER2 mutation. Note: A HER2 mutation documented only from a liquid biopsy samples cannot be used for enrollment.
* Had previous treatment including platinum therapy in the metastatic/locally advanced setting and not amenable to curative surgery or radiation. Participant must have progressed during or after the last treatment regimen or discontinued because of unacceptable toxicity.
* Presence of at least 1 measurable lesion confirmed by the blinded Independent Central Review based on RECIST version 1.1
* Willing and able to provide an archival tumor tissue sample. A fresh biopsy is required if an archival tumor tissue sample cannot be supplied. Resection and core needle biopsy are acceptable. Fine needle aspirates or cell block are not acceptable.
* Eastern Cooperative Oncology Group performance status 0 to 1
* Left ventricular ejection fraction ≥ 50% within 28 days before randomization Resection and core needle biopsy are acceptable - Adequate organ function as specified in protocol within 14 days before randomization
* Adequate treatment washout period before randomization
* Participants of reproductive/childbearing potential agree to use a highly effective form of contraception (or avoid intercourse) during study period and up to 7 months (females) and 4 months (males) after last study dose
* Males should not freeze or donate sperm throughout the study period up to at least 4 months after last study dose; females should not donate or retrieve ova for their own use throughout the study period and up to at least 7 months after last study dose
* Life expectancy 3 months or more

Exclusion Criteria:

* Known driver mutation in the epidermal growth factor receptor (EGFR), BRAF, or MET exon 14 gene or a known anaplastic lymphoma kinase (ALK), ROS1, RET, or NTRK fusion
* Medical history of myocardial infarction within 6 months before randomization, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV). Participants with troponin levels above upper limit of normal at screening (as defined by the manufacturer) and without any myocardial infarction (MI)-related symptoms should have a cardiologic consultation before randomization to rule out MI
* Corrected QT interval (QTcF) prolongation > 470 msec (females) or >450 msec (males) based on average of the triplicate12-lead electrocardiogram at screening
* History of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated
* History of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the participant's participation in the clinical study or evaluation of the clinical study results
* Known human immunodeficiency virus (HIV) infection
* Known active, clinically relevant liver disease (eg, active hepatitis B, or active hepatitis C) such as those with serologic evidence of viral infection within 28 days of Cycle 1, Day 1
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline
* Pregnant, breastfeeding, or planning to become pregnant
* Otherwise considered inappropriate for the study by the Investigator
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg. pulmonary emboli within three months of the study randomization, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.)
* Any autoimmune, connective tissue or inflammatory disorders (e.g., Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening
* Prior complete pneumonectomy
* Had prior treatment with any agent, including an antibody drug conjugate (ADC), containing a chemotherapeutic agent targeting topoisomerase I

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (50):
- United States (11):
  - University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital (MGH) - Hematology/Oncology, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute/Henry Ford Hospital, Detroit, Michigan
  - University of Michigan, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virgina Cancer Specialists, Fairfax, Virginia
- Australia (2):
  - St John of God Subiaco Hospital, Subiaco
  - Princess Alexandra Hospital, Woolloongabba
- University Health Network, Toronto, Canada
- France (6):
  - Centre Leon Berard, Lyon
  - Assistance Publique Hopitaux de Marseille AP-HM, Hopital NORD, Marseille
  - Hopital Pontchaillou, Rennes
  - CHU Nantes, Saint-Herblain
  - CHU toulouse - hÃ´pital Larrey, Toulouse
  - Gustav Roussy, Villejuif
- Italy (6):
  - Ospedale San Luca, Lucca
  - IRCCS Istituto Europeo di Oncologia, Milan
  - SC Oncologia, AOU Policlinico Modena, Modena
  - Istituto Nazionale Tumori Fondazione G. Pascale di Napoli Strutturadi Oncologia, Napoli
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Humanitas Cancer Center Istituto Clinico Humanitas, Rozzano
- Japan (6):
  - Aichi Cancer Center Hospital, Chikusa
  - National Cancer Central Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Ōsaka-sayama
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Erasmus MC, Rotterdam
- South Korea (5):
  - Chungbuk National University Hospital, Jungbuk
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Clinica Univ. de Navarra - P, Pamplona
  - Hospital Universitari i PolitÃ¨cnic La Fe, Valencia
- Taiwan (5):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital CGMH - LinKou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Janne PA, Goto Y, Kubo T, Ninomiya K, Kim SW, Planchard D, Ahn MJ, Smit E, Johannes de Langen A, Perol M, Pons-Tostivint E, Novello S, Hayashi H, Shimizu J, Kim DW, Pereira K, Cheng FC, Taguchi A, Cheng Y, Dunton K, Ali A, Goto K. Final Analysis Results and Patient-Reported Outcomes From DESTINY-Lung02-A Dose-Blinded, Randomized, Phase 2 Study of Trastuzumab Deruxtecan in Patients With HER2-Mutant Metastatic NSCLC. J Thorac Oncol. 2025 Dec;20(12):1814-1828. doi: 10.1016/j.jtho.2025.07.129. Epub 2025 Jul 30. PMID 40749900
- [Derived] Goto K, Goto Y, Kubo T, Ninomiya K, Kim SW, Planchard D, Ahn MJ, Smit EF, de Langen AJ, Perol M, Pons-Tostivint E, Novello S, Hayashi H, Shimizu J, Kim DW, Kuo CH, Yang JC, Pereira K, Cheng FC, Taguchi A, Cheng Y, Feng W, Tsuchihashi Z, Janne PA. Trastuzumab Deruxtecan in Patients With HER2-Mutant Metastatic Non-Small-Cell Lung Cancer: Primary Results From the Randomized, Phase II DESTINY-Lung02 Trial. J Clin Oncol. 2023 Nov 1;41(31):4852-4863. doi: 10.1200/JCO.23.01361. Epub 2023 Sep 11. PMID 37694347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 152 participants were enrolled and treated at clinic centers in North America, Europe, and Asia-Pacific.
Groups:
- Trastuzumab Deruxtecan 5.4 mg/kg: Participants randomized to receive trastuzumab deruxtecan 5.4 mg/kg, administered by intravenous infusion every 3 weeks (Q3W).
- Trastuzumab Deruxtecan 6.4 mg/kg: Participants randomized to receive trastuzumab deruxtecan 6.4 mg/kg, administered by intravenous infusion every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Started | 102 | 50
Completed | 0 | 0
Not Completed | 102 | 50
Not completed — Death | 4 | 2
Not completed — Adverse Event | 18 | 19
Not completed — Progressive Disease | 61 | 23
Not completed — Clinical Progression | 4 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 4 | 0
Not completed — Other | 6 | 3
Not completed — Randomized but not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg | Total
Number analyzed (Participants) | 102 | 50 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 35 | 97
  >=65 years | 40 | 15 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.59) | 59.5 (12.14) | 59.7 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 34 | 99
  Male | 37 | 16 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 65 | 31 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 23 | 5 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response Rate by Blinded Independent Central Review Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer
Description: Confirmed objective response rate (ORR), defined as the proportion of participants with complete response (CR) or partial response (PR), was assessed by blinded independent central review (BICR) based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: 9 months after the last participant is randomized to data cut off, up to approximately 21 months
Population: Full Analysis Set includes all subjects for whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
percentage of participants | 50.0 [39.9 to 60.1] | 56.0 [41.3 to 70.0]

2. Secondary Outcome: Percentage of Participants With Confirmed Objective Response Rate by Investigator Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung CancerTumors
Description: Confirmed objective response rate (ORR), defined as the percentage of participants with complete response (CR) or partial response (PR), will be assessed by the Investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Full Analysis Set includes all subjects for whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
Percentage of participants | 46.1 [36.2 to 56.2] | 56.0 [41.3 to 70.0]

3. Secondary Outcome: Duration of Response Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer
Description: Duration of response (DoR) is defined as the time from the initial response (complete response [CR] or partial response [PR]) until documented tumor progression or death from any cause. DoR is only defined for participants who achieved confirmed CR or PR. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Full Analysis Set includes all subjects for whom study treatment was assigned by randomization. From the Full Analysis Set, 47 participants had a confirmed CR or PR in T-DXd 5.4 mg/kg arm, and 28 participants in T-DXd 6.4 mg/kg arm
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 47 | 28
months | 11.1 [8.3 to 15.5] | 12.9 [6.9 to 15.4]

4. Secondary Outcome: Disease Control Rate Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer
Description: Disease control rate (DCR) is the sum of complete response (CR), partial response (PR), and stable disease (SD) rates. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Full Analysis Set includes all subjects for whom study treatment was assigned by randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
Percentage of participants | 90.2 [82.7 to 95.2] | 88.0 [75.7 to 95.5]

5. Secondary Outcome: Progression-free Survival Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer
Description: Progression-free survival (PFS) is defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on blinded independent central review (BICR) and investigator assessment.
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Full Analysis Set includes all subjects for whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
months | 9.7 [8.2 to 11.3] | 9.5 [6.5 to 15.1]

6. Secondary Outcome: Overall Survival Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer Tumors
Description: Overall survival (OS) is defined as the time from date of randomization until death from any cause.
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
months | 19.0 [14.7 to NA] — Not estimable due to insufficient number of participants with events | 17.9 [13.8 to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: The Percentage of Participants Reporting Treatment-emergent Adverse Events Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer Tumors
Time Frame: 9 months after the last participant is randomized or later to data cut off, up to approximately 35 months
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
Participants | 101 | 50

8. Secondary Outcome: Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) for Trastuzumab Deruxtecan, Total Anti-HER2 Antibody, and Active Metabolite MAAA-1181a
Time Frame: Cycle 1 Day 1; Cycle 2 Day 1, and Cycle 3 Day 1: pre- and post-dose; Cycle 1 Day 8: 7 days post-dose; Cycle 1 Day 15: 14 days post-dose; Cycle 4 Day 1 and Cycle 6 Day 1: pre-dose (each cycle is 21 days)
Population: The PK Analysis Set included all randomized subjects who received at least one dose of study drug and had any measurable post-dose serum concentrations of T-DXd, total anti-HER2 antibody, and DXd.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 101 | 50
µg/mL
  Trastuzumab Deruxtecan | 148 (69.5) | 196 (184)
  Total Anti-HER2 Antibody | 138 (57.8) | 179 (194)
  DXd (Metabolite Active Metabolite MAAA-1181a) | .015 (.007) | .018 (.008)

9. Secondary Outcome: Pharmacokinetic Parameter Minimum Observed Concentration (Ctrough) for Trastuzumab Deruxtecan, Total Anti-HER2 Antibody, and Active Metabolite MAAA-1181a
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 101 | 50
µg/mL
  Trastuzumab Deruxtecan | 5.47 (11.1) | 5.84 (3.48)
  Total Anti-HER2 Antibody | 6.39 (10.7) | 7.16 (5.00)
  DXd (Metabolite Active Metabolite MAAA-1181a) | .0003 (.0003) | .0003 (.0002)

10. Secondary Outcome: Pharmacokinetic Parameter Area Under the Serum Concentration-Time Curve (AUC) for Trastuzumab Deruxtecan, Total Anti-HER2 Antibody, and Active Metabolite MAAA-1181a
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: µg × d/mL
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 101 | 50
µg × d/mL
  Trastuzumab Deruxtecan | 658 (185) | 793 (210)
  Total Anti-HER2 Antibody | 697 (208) | 829 (261)
  DXd (Metabolite Active Metabolite MAAA-1181a) | .050 (.022) | .059 (.017)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Following Intravenous Administration of Trastuzumab Deruxtecan in Participants With Metastatic Non-small Cell Lung Cancer Tumors
Time Frame: Pre-dose on Day 1 of Cycles 1, 2 and 4, and then every 4 cycles (each cycle is 21 days), up to Cycle 28 and End of Treatment.
Population: The Immunogenicity Analysis Set included all subjects who received at least one dose of the study drug and who had at least one baseline or post-baseline immunogenicity assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 101 | 50
Participants | 2 | 1

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) and EORTC Quality of Life Questionnaire for Lung Cancer Trials (QLQ-LC13) Scores
Description: The EORTC QLQ-C30 consists of 30 questions assessing global health-related quality of life, five aspects of subject functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), and six single-items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. Higher scores for functioning scales and global health status indicate a better level of functioning while higher scores on the symptom and single-item scales indicate a higher level of symptoms. The QLQ-LC13 is a 13-item questionnaire designed to assess lung cancer-related symptoms and treatment side effects. The scales ranges from 1=not at all to 4=very much. The summation of scores range from 0 to 100, where higher scores represent increasing symptoms levels.
  scales.
Time Frame: At baseline and at end of treatment 40-day follow-up visit
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
score on scale
  QLQ-C30: Change from Baseline 40-Day Follow-up | -1.11 (17.780) | 15.63 (31.947)
  QLQ-LC13: Change from Baseline 40-Day Follow-up | -2.38 (24.335) | -29.17 (27.817)

13. Secondary Outcome: Time to Deterioration in European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) Scores
Description: The EORTC QLQ-C30 consists of 30 questions assessing global health-related quality of life, five aspects of subject functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), and six single-items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. Higher scores for functioning scales and global health status indicate a better level of functioning while higher scores on the symptom and single-item scales indicate a higher level of symptoms.
Time Frame: At baseline and at end of treatment 40-day follow-up visit
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
Number analyzed (Participants) | 102 | 50
months | 8.6 [4.9 to 11.4] | 9.3 [2.5 to NA] — Not estimable due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug, up to approximately 35 months
Description: A treatment-emergent adverse event (TEAE) was defined as an AE that occurred, having been absent before the first dose of study drug, or had worsened after initiating study treatment up until 47 days after the last dose of the study treatment. All-Cause Mortality was assessed in the Full Analysis Set, all adverse events were assessed in the Safety Analysis Set
Arm/Group | Trastuzumab Deruxtecan 5.4 mg/kg | Trastuzumab Deruxtecan 6.4 mg/kg
All-Cause Mortality (participants affected / at risk) | 52/102 | 24/50
Serious Adverse Events (participants affected / at risk) | 42/101 | 26/50
Other Adverse Events (participants affected / at risk) | 101/101 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Deruxtecan 5.4 mg/kg (N=101) | Trastuzumab Deruxtecan 6.4 mg/kg (N=50)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (4)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Deruxtecan 5.4 mg/kg (N=101) | Trastuzumab Deruxtecan 6.4 mg/kg (N=50)
Anaemia (Blood and lymphatic system disorders) | 41 (113) | 24 (81)
Neutropenia (Blood and lymphatic system disorders) | 13 (35) | 8 (29)
Nausea (Gastrointestinal disorders) | 69 (166) | 41 (85)
Constipation (Gastrointestinal disorders) | 38 (56) | 17 (26)
Vomiting (Gastrointestinal disorders) | 31 (63) | 22 (38)
Diarrhoea (Gastrointestinal disorders) | 25 (42) | 18 (32)
Stomatitis (Gastrointestinal disorders) | 15 (22) | 7 (12)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 7 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 3 (5) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3)
Asthenia (General disorders) | 19 (46) | 13 (42)
Fatigue (General disorders) | 16 (18) | 7 (16)
Malaise (General disorders) | 16 (43) | 5 (8)
Pyrexia (General disorders) | 12 (18) | 8 (10)
Oedema peripheral (General disorders) | 4 (5) | 3 (4)
Chest pain (General disorders) | 3 (3) | 4 (6)
COVID-19 (Infections and infestations) | 17 (21) | 9 (11)
Paronychia (Infections and infestations) | 8 (11) | 1 (1)
Pneumonia (Infections and infestations) | 7 (9) | 7 (10)
Urinary tract infection (Infections and infestations) | 4 (7) | 5 (5)
Neutrophil count decreased (Investigations) | 32 (171) | 20 (79)
White blood cell count decreased (Infections and infestations) | 26 (118) | 16 (68)
Platelet count decreased (Investigations) | 26 (118) | 16 (68)
Aspartate aminotransferase increased (Investigations) | 21 (36) | 7 (17)
Alanine aminotransferase increased (Investigations) | 14 (28) | 8 (13)
Weight decreased (Investigations) | 17 (32) | 7 (7)
Blood creatinine increased (Investigations) | 6 (8) | 4 (5)
Blood bilirubin increased (Investigations) | 3 (12) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 41 (64) | 25 (49)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (26) | 3 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 13 (17) | 1 (2)
Headache (Nervous system disorders) | 7 (7) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 7 (7)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (26) | 17 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (15) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (17) | 3 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04644237/Prot_SAP_000.pdf